CLINICAL TRIAL: NCT00339456
Title: A Randomized, Controlled Trial of Short Cycle Intermittent Versus Continuous HAART for the Treatment of Chronic HIV Infection in Uganda
Brief Title: Intermittent Versus Continuous HAART (Highly Active Antiretroviral Therapy) for Treating Chronic HIV Infected Patients in Uganda
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999902288; 02-I-N288
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-05-20

CONDITIONS: HIV
Keywords: Therapy; Africa; Structured; Interruption; Antiretroviral; HIV
MeSH Terms: interventions — Antiretroviral Therapy, Highly Active

INTERVENTIONS:
Drug: HAART

SUMMARY:
Although highly active antiretroviral therapy (HAART) has been successful in suppressing plasma HIV RNA levels and providing significant clinical benefit in infected patients, it does not eradicate HIV infection. It is now clear that virus replication persists despite undetectable plasma viremia in individuals receiving HAART. In this regard, withdrawing HAART, even after prolonged periods of virus suppression, leads almost invariably to a rapid rebound of plasma viremia. It is also now clear that prolonged, continuous HAART carries a risk of significant toxicity and side effects. In addition, the monetary cost of HAART is prohibitive for many individuals and countries. In terms of cost, 95% of the HIV-infected individuals in the world are beyond the reach of therapy as a direct consequence of the cost of therapy. These observations may argue for a different approach to HAART with the goals of: 1) durable suppression of virus replication, without an attempt at eradication, 2) minimization of toxicity and side effects and improvement in patient life-style, and 3) a reduction in cost. Preliminary data from a pilot study conducted at the National Institutes of Allergy and Infectious Diseases, USA, have demonstrated that short cycle structured intermittent therapy, 7 days HAART drug followed by 7 days off HAART has maintained suppression of plasma HIV RNA while preserving CD4+ T cell counts for up to 80 weeks. In addition, there was no evidence for increased HIV in reservoir sites; nor was there evidence for the development of resistance to antiretroviral drugs. Finally, there was a decrease in parameters of toxicity. This approach may have particular applicability for the treatment of HIV in the Southern Hemisphere. Therefore, we propose to study the virologic and immunologic effects of short cycle intermittent versus continuous HAART in HIV-infected individuals from the JCRC (Kampala, Uganda) in a randomized, controlled, intent-to-treat trial. We shall evaluate both the 7 days on-HAART/7 days off-HAART as well as a 2 days off-HAART/5 days on-HAART approach. In December, 2004, the 7/7 arm was discontinued....

DETAILED DESCRIPTION:
Although highly active antiretroviral therapy (HAART) has been successful in suppressing plasma HIV RNA levels and providing significant clinical benefit in infected patients, it does not eradicate HIV infection. It is now clear that virus replication persists despite undetectable plasma viremia in individuals receiving HAART. In this regard, withdrawing HAART, even after prolonged periods of virus suppression, leads almost invariably to a rapid rebound of plasma viremia. It is also now clear that prolonged, continuous HAART carries a risk of significant toxicity and side effects. In addition, the monetary cost of HAART is prohibitive for many individuals and countries. In terms of cost, 95 percent of the HIV-infected individuals in the world are beyond the reach of therapy as a direct consequence of the cost of therapy. These observations may argue for a different approach to HAART with the goals of: 1) durable suppression of virus replication, without an attempt at eradication, 2) minimization of toxicity and side effects and improvement in patient life-style, and 3) a reduction in cost. Preliminary data from a pilot study conducted at the National Institutes of Allergy and Infectious Diseases, USA, have demonstrated that short cycle structured intermittent therapy, 7 days HAART drug followed by 7 days off HAART has maintained suppression of plasma HIV RNA while preserving CD4+ T cell counts for up to 80 weeks. In addition, there was no evidence for increased HIV in reservoir sites; nor was there evidence for the development of resistance to antiretroviral drugs. Finally, there was a decrease in parameters of toxicity. This approach may have particular applicability for the treatment of HIV in the Southern Hemisphere. Therefore, we propose to study the virologic and immunologic effects of short cycle intermittent versus continuous HAART in HIV-infected individuals from the JCRC (Kampala, Uganda) in a randomized, controlled, intent-to-treat trial. We shall evaluate both the 7 days on-HAART/7 days off-HAART as well as a 2 days off-HAART/5 days on-HAART approach. In December, 2004, the 7/7 arm was discontinued.

ELIGIBILITY:
* INCLUSION CRITERIA:

Documentation of HIV-1 infection by licensed ELISA test kit and confirmed by a second method (e.g. Western Blot).

Absolute CD4+ T-cell count of greater than or equal to 125/mm(3) within 30 days before randomization (For patients who are status post-splenectomy, also CD4+ T-cell greater than 20%).

If the CD4+ T cell count is less than or equal to 200 cells/mm(3), the patient must be receiving PCP prophylaxis.

Receiving at least 3-drug HAART with the most recent viral load test prior to screening less than 500 copies/ml. Patients must be receiving 3 drug HAART containing an NNRTI, abacavir or PI for at least 90 days prior to enrollment and at least 1 PI or efavirenz for 30 days prior to enrollment.

A viral load of less than 50 copies/ml prior to enrollment.

Age at least 18 years and above.

For women of childbearing potential, a negative pregnancy test (serum or urine) is required within 14 days prior to randomization.

Laboratory values (within 30 days prior to randomization):

1. AST no more than 5 X the upper limit of normal (ULN).
2. Total or direct bilirubin no more than 2 X ULN unless there is a pattern consistent with Gilbert s syndrome or the patient is receiving indinavir.
3. Creatinine no more than 2.0 mg/dL.
4. Platelet count at least 50,000/microliters.

Written consent to participate in the trial.

Patient financially capable of purchasing the drugs uninterrupted for at least 72 weeks (the duration of the study).

EXCLUSION CRITERIA:

Concurrent malignancy, or any other disease state, requiring cytotoxic chemotherapy.

Symptomatic for significant HIV-related illnesses, such as opportunistic infections and malignancies other than mucocutaneous Kaposi s sarcoma. A history of AIDS defining opportunistic infections other than mucocutaneous Kaposi s sarcoma or candida or treated tuberculosis.

Use of experimental antiretroviral less than or equal to 6 months prior to enrollment. An exception may be made for hydroxeurea according to the judgment of the Principal Investigator.

Pregnancy or breastfeeding.

Significant cardiac, pulmonary, kidney, rheumatologic, gastrointestinal, or CNS disease as detectable on routine history, physical examination, or screening laboratory studies. If an abnormality is a contraindication to a specific drug, an alternative drug within the same class may be used.

Psychiatric illness that, in the opinion of the PI, might interfere with study compliance.

Active substance abuse or history of prior substance abuse that may interfere with protocol compliance or compromise patient safety.

Refusal to practice safe sex or use precautions against pregnancy (effective birth control with barrier contraceptives or abstinence).

Known history or laboratory evidence of chronic hepatitis B infection including surface antigen positivity.

Receiving salvage HAART, i.e. evidence of clinical resistance to licensed anti-retrovirals as indicated by clinical progression, an elevated viral load or declining CD4+ T cell count while receiving antiretroviral therapy, or receiving sub-optimal antiretroviral therapy prior to HAART.

Patients currently receiving nevirapine or abacavir are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2002-08-21; Primary Completion 2008-02-01 (Actual); Study Completion 2008-02-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of short cycle intermittent versus continuous HAART on viral load.

SECONDARY OUTCOMES:
To evaluate change in CD4 T-cell counts, change in virus patterns, toxicity and side effects, Quality of Life, and adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Quinn, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Joint Clinical Research Center, Kampala, Uganda

REFERENCES:
- [Background] Natarajan V, Bosche M, Metcalf JA, Ward DJ, Lane HC, Kovacs JA. HIV-1 replication in patients with undetectable plasma virus receiving HAART. Highly active antiretroviral therapy. Lancet. 1999 Jan 9;353(9147):119-20. doi: 10.1016/s0140-6736(05)76156-0. No abstract available. PMID 10023903
- [Background] Furtado MR, Callaway DS, Phair JP, Kunstman KJ, Stanton JL, Macken CA, Perelson AS, Wolinsky SM. Persistence of HIV-1 transcription in peripheral-blood mononuclear cells in patients receiving potent antiretroviral therapy. N Engl J Med. 1999 May 27;340(21):1614-22. doi: 10.1056/NEJM199905273402102. PMID 10341273
- [Background] Zhang L, Ramratnam B, Tenner-Racz K, He Y, Vesanen M, Lewin S, Talal A, Racz P, Perelson AS, Korber BT, Markowitz M, Ho DD. Quantifying residual HIV-1 replication in patients receiving combination antiretroviral therapy. N Engl J Med. 1999 May 27;340(21):1605-13. doi: 10.1056/NEJM199905273402101. PMID 10341272
- [Derived] Reynolds SJ, Kityo C, Hallahan CW, Kabuye G, Atwiine D, Mbamanya F, Ssali F, Dewar R, Daucher M, Davey RT Jr, Mugyenyi P, Fauci AS, Quinn TC, Dybul MR. A randomized, controlled, trial of short cycle intermittent compared to continuous antiretroviral therapy for the treatment of HIV infection in Uganda. PLoS One. 2010 Apr 22;5(4):e10307. doi: 10.1371/journal.pone.0010307. PMID 20442758